CLINICAL TRIAL: NCT03006094
Title: Validity, Reliability and Responsiveness of the Greek Version of the Chronic Pain Grade Questionnaire (CPGQ) in Chronic Hip Pain Sufferers
Brief Title: The Greek Version of the Chronic Pain Grade Questionnaire (CPGQ)
Status: Completed | Type: Observational
Sponsor: Asklepieion Voulas General Hospital (Other Government)
Responsible Party: Principal Investigator, Maria Diakomi, MD, MSc, Asklepieion Voulas General Hospital
Other Study IDs: 242
Record Dates: First submitted 2016-12-22; First posted 2016-12-30 (Estimated); Last update posted 2018-03-06 (Actual); Status verified 2018-03

CONDITIONS: Chronic Hip Pain
Keywords: questionnaire; hip; pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the present study is to investigate and report on the psychometric properties of a Greek version of the Chronic Pain Grade Questionnaire (CPGQ).

DETAILED DESCRIPTION:
The Chronic Pain Grade Questionnaire (CPGQ) is designed to evaluate overall severity of chronic pain based on two dimensions, pain intensity and pain-related disability. Currently, there is no reliable, valid and sensitive to change self-report instrument as brief and easy to understand and complete as the CPGQ available in Greek. A culturally adapted version of the CPGQ would facilitate the study of chronic pain and its implications in the Greek population and allow for cross-cultural comparisons. The aim of the present study is to examine the validity, reliability and responsiveness of a Greek version of the CPGQ in chronic hip pain sufferers.

ELIGIBILITY:
Inclusion Criteria:

* chronic hip pain (persistent or recurrent hip pain for at least 12 weeks)

Exclusion Criteria:

* severe systemic disease that is a constant threat to life
* known psychiatric disorder
* impaired cognition or dementia
* mother language other than Greek

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Orthopaedic outpatients
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Factor analysis of the Greek version of the CPGQ | At recruitment (baseline)
Correlations between the CPGQ items, total, subscale scores and the SF-12 PCS, MCS scores | At recruitment (baseline)
Cronbach's alpha values for the total scale and each subscale of the Greek version of the CPGQ | At recruitment (baseline)
Intraclass correlation coefficient (ICC) values for the total scale and each sub scale of the Greek version of the CPGQ | 48 hours
Change in CPGQ total scale and subscale scores | At recruitment (baseline) and 6 months following total hip replacement surgery
  Recruited subjects who will undergo total hip replacement surgery will complete the Greek version of the CPGQ and report their improvement using a dichotomous variable (Yes or No improvement) six months postoperatively.

SECONDARY OUTCOMES:
Percentage of patients who were able to complete the Greek version of the CPGQ by themselves | At recruitment (baseline)
Time employed in filling out the Greek version of the CPGQ | At recruitment (baseline)

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital Asklepieio Voulas, Voula, Greece

IPD SHARING:
Plan to Share IPD: No